CLINICAL TRIAL: NCT01815177
Title: Advantages of Arthroscopic Rotator Cuff Repair With Transosseous Suture Technique. A Prospective Randomized Controlled Trial
Brief Title: Arthroscopic Rotator Cuff Repair: Suture Anchors Versus Arthroscopic Transosseous Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Pietro Randelli, MD, Assistant Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shoulder01
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Suture Anchors

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthroscopic transosseous fixation (Experimental): Patients with torn rotator cuff randomized to experimental treatment receive a complete arthroscopic transosseous cuff repair
  Interventions: Device: Arthroscopic transosseous fixation
- Repair using suture anchors (Other): Patients randomized to this arm receive an arthroscopic rotator cuff repair using suture anchors.
  Interventions: Device: Suture anchors

INTERVENTIONS:
Device: Arthroscopic transosseous fixation
  Other Names: ArthroTunneler transosseous tunneling device (Tornier Inc)
  Arms: Arthroscopic transosseous fixation
Device: Suture anchors
  Arms: Repair using suture anchors

SUMMARY:
Arthroscopic transosseous fixation of rotator cuff tears has become an alternative to arthroscopic suture anchor.

This novel technique that allows surgeons to perform a standardized arthroscopic transosseous (anchor free) repair of rotator cuff tears can improve postoperative pain and reduce the incidence of shoulder stiffness.

The aim of the this study is to compare clinical outcomes of two groups of patients: patients that received an arthroscopic transosseous fixation using the ArthroTunneler tunneling device (Tornier Inc, Edina, Minnesota) versus patients that received an arthroscopic rotator cuff repair using suture anchors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18, <65
* Rotator cuff tears
* Patients given written informed consent
* BMI ≤ 33

Exclusion Criteria:

* Age > 65, < 18
* previous surgical intervention
* Informed consent not accepted
* Serious comorbidity
* Diabetes
* Metabolic Disorders
* Active infections
* Muscular Atrophy
* Biceps Tenodesis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pain | first 28 days after surgery
  Paracetamol/Codeine 500/30 is given to every patient at 08.00 and 20.00 for the first 5 days. The patient is highly recommended to indicate his pain at 19.30 and to write if there is any modification in the assumption of pain killers.

SECONDARY OUTCOMES:
Shoulder Stiffness | Postoperative passive range of motion is measured 2 months after surgery
  For evaluation of shoulder stiffness, passive range of motion is measured with a goniometer by a single examiner in 3 directions: forward elevation, external rotation at the side and internal rotation at the back

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Randelli, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- Policlinico San Donato (istituto di ricovero e cura a carattere scientifico), San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garofalo R, Castagna A, Borroni M, Krishnan SG. Arthroscopic transosseous (anchorless) rotator cuff repair. Knee Surg Sports Traumatol Arthrosc. 2012 Jun;20(6):1031-5. doi: 10.1007/s00167-011-1725-4. Epub 2011 Oct 20. PMID 22011882
- [Background] Voos JE, Barnthouse CD, Scott AR. Arthroscopic rotator cuff repair: techniques in 2012. Clin Sports Med. 2012 Oct;31(4):633-44. doi: 10.1016/j.csm.2012.07.002. PMID 23040550
- [Background] Longo UG, Franceschi F, Berton A, Maffulli N, Denaro V. Arthroscopic transosseous rotator cuff repair. Med Sport Sci. 2012;57:142-152. doi: 10.1159/000328900. Epub 2011 Oct 4. PMID 21986052
- [Background] Salata MJ, Sherman SL, Lin EC, Sershon RA, Gupta A, Shewman E, Wang VM, Cole BJ, Romeo AA, Verma NN. Biomechanical evaluation of transosseous rotator cuff repair: do anchors really matter? Am J Sports Med. 2013 Feb;41(2):283-90. doi: 10.1177/0363546512469092. Epub 2012 Dec 13. PMID 23239668
- [Background] Garrigues GE, Lazarus MD. Arthroscopic bone tunnel augmentation for rotator cuff repair. Orthopedics. 2012 May;35(5):392-7. doi: 10.3928/01477447-20120426-04. PMID 22588393
- [Derived] Randelli P, Stoppani CA, Zaolino C, Menon A, Randelli F, Cabitza P. Advantages of Arthroscopic Rotator Cuff Repair With a Transosseous Suture Technique: A Prospective Randomized Controlled Trial. Am J Sports Med. 2017 Jul;45(9):2000-2009. doi: 10.1177/0363546517695789. Epub 2017 Mar 24. PMID 28339286